CLINICAL TRIAL: NCT01003249
Title: Treatment of Patients With Dysfunctional Voiding and Lower Urinary Tract Symptoms With Baclofen: a Randomized Double-blind Placebo-controlled Cross-over Trial
Brief Title: Dysfunctional Voiding and Lower Urinary Tract Symptoms With Baclofen
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment was going too slowly
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00009516
Record Dates: First submitted 2009-10-21; First posted 2009-10-28 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Overactive Bladder; Constipation; Lower Urinary Tract Symptoms
Keywords: over distention of bladder; Dysfunctional voiding; dysfunctional elimination syndrome
MeSH Terms: conditions — Urinary Bladder, Overactive; Constipation; Lower Urinary Tract Symptoms | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baclofen, Then Placebo (Active Comparator): Subjects will then randomly be assigned in placebo or baclofen groups. Daily dose will be doubled every three days, up to 80 mg or when side effects appear. There will be a washout period after three week. At the end of 4 week drug will be tapered (halved every 2 days and quitted after 2 days of using 20 mg baclofen). Then patients initially assigned to the baclofen group will be assigned to the placebo group, and those assigned to the placebo group will be assigned to the baclofen group. Patients would then receive a dose of baclofen 10 mg PO twice daily (or placebo twice daily), and then the dose will be escalated to 80 mg
  Interventions: Drug: Baclofen; Drug: Placebo
- Placebo, Then Baclofen (Placebo Comparator): Subjects will then randomly be assigned in placebo or baclofen groups. Daily dose will be doubled every three days, up to 80 mg or when side effects appear. There will be a washout period after three week. At the end of 4 week drug will be tapered (halved every 2 days and quitted after 2 days of using 20 mg baclofen). Then patients initially assigned to the baclofen group will be assigned to the placebo group, and those assigned to the placebo group will be assigned to the baclofen group. Patients would then receive a dose of baclofen 10 mg PO twice daily (or placebo twice daily), and then the dose will be escalated to 80 mg
  Interventions: Drug: Baclofen; Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — Subjects will be randomly assigned to placebo or baclofen groups. Daily dose will be doubled every three days, up to 80 mg or when side effects appear. At the end of 4 week drug will be tapered (halved every 2 days and quitted after 2 days of using 20 mg baclofen). After the 3 week washout period, questionnaires, diary, EMG and uroflowmetry will be repeated. Then patients initially assigned to the baclofen group will be assigned to the placebo group, and those assigned to the placebo group will be assigned to the baclofen group.
  Patients would then receive a dose of baclofen 10 mg PO twice daily (or placebo twice daily), and then the dose will be escalated to 80 mg.
Drug: Placebo — Subjects will then randomly be assigned in placebo or baclofen groups. Daily dose will be doubled every three days, up to 80 mg or when side effects appear. At the end of 4 week drug will be tapered (halved every 2 days and quitted after 2 days of using 20 mg baclofen). After the 3 week washout period, questionnaires, diary, EMG and uroflowmetry will be repeated. Then patients initially assigned to the baclofen group will be assigned to the placebo group, and those assigned to the placebo group will be assigned to the baclofen group.
  Patients would then receive a dose of baclofen 10 mg PO twice daily (or placebo twice daily), and then the dose will be escalated to 80 mg.

SUMMARY:
Dysfunctional voiding is often associated with constipation. The association of constipation with urologic pathologic processes has previously been described since the 1950's, but it was only over the past decade that clinicians have paid more attention to this relationship and recognized it existence with the term dysfunctional elimination syndrome (DES). This term is used to reflect the broad spectrum of functional disturbances that may affect the urinary tract including that of functional bowl disturbances and can be classified as follows:

* Functional disorder of filling: overactive bladder, over distention of bladder or insensate bladder, which may be associated with fecal impaction or rectal distention with infrequent bowel movements
* Functional disorder of emptying: over-recruitment of pelvic floor activity during voiding causing interrupted and/or incomplete emptying also associated with defecation difficulties due to non- relaxation of the puborectalis muscle, dyssynergic defecation or pain with defecation Several different therapeutic options have been used for patients with dysfunctional voiding mainly to decrease bladder outlet obstruction. These treatments including, alpha adrenergic antagonists, and botulinum toxin are less than optimum. One possible explanation for these drug failures includes the inability of these medications to relax the striated muscles of the pelvic floor necessary for voiding.

To date there has been no data to evaluate the role of baclofen on the striated muscle of the external anal sphincter, essential in the defecation process.

DETAILED DESCRIPTION:
Outcome Measure(s)

1. Efficacy of baclofen vs. placebo on dysfunctional voiding as measured with uroflometry and EMG; patients' symptoms score questionnaires and diaries.
2. Efficacy of baclofen vs. placebo on the external anal sphincter muscle dysfunction via patient symptoms and questionnaire.

3. The safety of baclofen in patients with dysfunctional voiding (urinary and defecatory).

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women (>18 years old, <65 years old)
* Patients with lower urinary tract symptoms (hesitancy, intermittency decreased force and caliber of urinary stream, urgency, incontinence) and urodynamic finding compatible with diagnosis of DV in multichannel videourodynamics. (Non relaxation or over stimulation of EMG activity, and stress pattern of voiding)
* Established symptoms for at least six months
* Patients with defecatory symptom should have symptoms of constipation (must include 2 or more of the following: straining during 25% of defecations, hard or lumpy stools during 25% of defecation, sensation of incomplete evacuation upon defecations, sensation of anorectal blockage or obstruction during 25% of defecations, manual maneuvers to facilitate 25% of defecations; loose stools that are rarely present without the use of laxatives; insufficient criteria to meet the definition of IBS-C.

Exclusion Criteria:

* Overt neurogenic disease
* Significant bladder outlet obstruction
* Detrusor instability on Urodynamic study
* Detrusor hypo contractility due to neurogenic causes
* Previous pelvic radiation
* Present (and past) malignancy of bladder or prostate
* Present or recurrent UTI (3 or more documented UTI in the past year )
* Interstitial Cystitis
* Diabetic neuropathy
* Patients on anticholinergic medications
* Bladder stones
* Urinary retention
* Underlying dementia or significant cognitive impairment.
* Patients unwilling to undergo videourodynamic , EMG or anorectal manometry testing
* Sample size: 62 patients in total (calculation basis described on Statistical Plan for Data Analysis)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gopal Badlani, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Baclofen, Then Placebo: Participants first received Baclofen for a total of 2 weeks (beginning dose=10mg and dose escalated up to 80 mg as symptoms appear), and were then tapered off of Baclofen for 2 weeks (total time= 4 weeks). This was followed by a 3 week washout period and then 4 weeks of Placebo.
- Placebo, Then Baclofen: Participants received Placebo for 4 weeks, followed by a 3 week washout period. Participants then received Baclofen for a total of 2 weeks (beginning dose=10mg and dose escalated up to 80 mg as symptoms appear), and were then tapered off of Baclofen for 2 weeks (total time= 4 weeks).
Period: First Intervention (4 Weeks)
Arm/Group | Baclofen, Then Placebo | Placebo, Then Baclofen
Started | 7 | 5
Received Intervention | 7 | 5
Completed | 5 | 3
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Non-Serious Event | 1 | 1
Period: Washout (3 Weeks)
Arm/Group | Baclofen, Then Placebo | Placebo, Then Baclofen
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Baclofen, Then Placebo | Placebo, Then Baclofen
Started | 4 | 3
Completed | 3 | 2
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Includes all participants in the study. Participants were randomized to either study drug or placebo
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
  Unknown | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Urine Flow Rate, as Measured With Uroflometry
Description: Uroflometry with patch electrodes will also be completed at the end of this four week period. Higher flow rate denotes better outcome.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: ml/s
Groups:
- Baclofen: Subjects will then randomly be assigned in placebo or baclofen groups. Daily dose will be doubled every three days, up to 80 mg or when side effects appear. At the end of 4 week drug will be tapered (halved every 2 days and quitted after 2 days of using 20 mg baclofen).
  Baclofen: Subjects will be randomly assigned to placebo or baclofen groups. Daily dose will be doubled every three days, up to 80 mg or when side effects appear. At the end of 4 week drug will be tapered (halved every 2 days and quitted after 2 days of using 20 mg baclofen).
- Placebo: Subjects will then randomly be assigned in placebo or baclofen groups. Daily dose will be doubled every three days, up to 80 mg or when side effects appear. At the end of 4 week drug will be tapered (halved every 2 days and quitted after 2 days of using 20 mg baclofen).
  Placebo Comparator: Placebo: Subjects will then randomly be assigned in placebo or baclofen groups. Daily dose will be doubled every three days, up to 80 mg or when side effects appear. At the end of 4 week drug will be tapered (halved every 2 days and quitted after 2 days of using 20 mg baclofen).
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 12 | 12
ml/s
  Baseline | 7.9 (1.93) | 8.4 (1.7)
  After Treatment | 10.1 (3.01) | 8.9 (2.05)

2. Primary Outcome: Number of Participants Exhibiting Abnormal EMG Activity During Voiding
Description: EMG with patch electrodes was completed at the end of this four week period. The number of participants with EMG activity during voiding was collected. EMG activity during the voiding is considered abnormal and is a criteria for voiding dysfunction.Lower numbers denotes better outcomes.
Time Frame: Baseline and 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Baclofen: Baclofen: Subjects will be randomly assigned to placebo or baclofen groups. Daily dose will be doubled every three days, up to 80 mg or when side effects appear. At the end of 4 week drug will be tapered (halved every 2 days and quitted after 2 days of using 20 mg baclofen).
- Placebo: Placebo Comparator: Placebo: Subjects will then randomly be assigned in placebo or baclofen groups. Daily dose will be doubled every three days, up to 80 mg or when side effects appear. At the end of 4 week drug will be tapered (halved every 2 days and quitted after 2 days of using 20 mg baclofen).
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Baseline | 6 | 6
  After Treatment | 4 | 6

3. Primary Outcome: Average Scores on International Consultation on Incontinence Modular Questionnaire- Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol)
Description: Diagnosis of dysfunctional bladder is based on symptoms demonstrating no relaxation or over stimulation of external urinary sphincter during voiding. Symptoms will be scored by International Consultation on Incontinence Modular Questionnaire- Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol). The ICIQ-LUTSqol is a patient-completed questionnaire for evaluating quality of life (QoL) in urinary incontinent patients There are 20 items and the score range is 10-200. Higher scores denotes better outcomes.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 12 | 12
scores on a scale
  Baseline | 165.3 (13.2) | 174 (18.1)
  After Treatment | 120.7 (14.8) | 160 (15.8)

4. Primary Outcome: Average Scores on Dysfunctional Voiding as Measured With Quality of Life (QOL) Questionnaire
Description: This was measured using the Urogenital Distress Inventory (UDI-6). The UDI-6 is a symptom inventory specific to lower urinary tract dysfunction and genital prolapse. There are 6 items scored. The score range is from 0-100 Lower scores denotes better outcomes.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 12 | 12
scores on a scale
  Baseline | 15.1 (3.23) | 14.3 (3.70)
  After Treatment | 14.3 (2.56) | 12.8 (3.25)

5. Secondary Outcome: Number (and Percentage) of Participants With External Anal Sphincter Muscle Dysfunction Via Patient Symptoms.
Description: The percent of patient in each group who had defecation problem
Time Frame: Baseline and 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Baclofen: Subjects will be randomly assigned to placebo or baclofen groups. Daily dose will be doubled every three days, up to 80 mg or when side effects appear. At the end of 4 week drug will be tapered (halved every 2 days and quitted after 2 days of using 20 mg baclofen).
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Before Treatment | 4 | 3
  After Treatment | 2 | 3

6. Secondary Outcome: Efficacy of Baclofen vs. Placebo on Number of Voidings Per Day
Description: The number of voiding per day before and after treatment.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Baclofen | Placebo
Number analyzed (Participants) | 12 | 12
number of voids
  Baseline | 10.7 (2.93) | 10.3 (2.85)
  After Treatment | 8.3 (1.98) | 9.2 (2.27)

ADVERSE EVENTS:
Arm/Group | Baclofen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen (N=12) | Placebo (N=12)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) — flare up in psychosis history of subject
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen (N=12) | Placebo (N=12)
GI Symptoms (Gastrointestinal disorders) | 1 (1) | 1 (1) — Common GI symptoms: bloating, upset stomach, nausea, etc..All GI Symptoms were collected/recorded under a single adverse event term
Excessive Sleepiness (General disorders) | 1 (1) | 2 (2)
Feeling too loose (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes